CLINICAL TRIAL: NCT04760912
Title: Comparison of General Anesthesia With Use of Muscle Relaxation and General Anesthesia Without Muscle Relaxation on Recovery of Muscle Strength of the Patients
Brief Title: General Anesthesia With and Without Muscle Relaxation and Muscle Strength Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Martina Miklic Bublic, MD, PhD, Principal investigator, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 022
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Rocuronium; Muscle Weakness; General Anaesthesia
Keywords: Rocuronium; Muscle strength; Residual blockade
MeSH Terms: conditions — Muscle Weakness | interventions — Rocuronium; Anesthesia, General; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group general anesthesia without rocuronium (Experimental): 30 patient ASA classification 1-2 for general anesthesia. Standard anesthesia monitoring. After induction with Propofol and Sufentanil ( doses adjusted according to weight and age) anesthesia was maintained with sevorane. Muscle strength measured on three occasions with Yamar dinamometar for hand grip strength, before induciran to anesthesia and immediate after Salingeru from anesthesia, then again measured in first 24 hours.
  Interventions: Procedure: General anesthesia for surgery
- Active comparator: general anesthesia with rocuronium (Active Comparator): 30 patient ASA classification 1-2 for general anesthesia. Standard anesthesia monitoring with train-of-four (TOF). After induction with Propofol and Sufentanil (doses adjusted according to weight and age) and rocuronium 0,6 mg per kg, anesthesia maintained with sevorane. Muscle strength neasured with Yamar dinamometar for hand grip strength before induction to anesthesia and immediate after awakening from anesthesia, then again measured in first 24 hours.
  Interventions: Drug: Rocuronium; Procedure: General anesthesia for surgery

INTERVENTIONS:
Drug: Rocuronium — Rocuronium used for neuromuscular blokade during anesthesia and anesthesia without rocuronium
  Other Names: Rocuronium bromide
  Arms: Active comparator: general anesthesia with rocuronium
Procedure: General anesthesia for surgery — General anesthesia with standard anesthetic monitoring,
  Other Names: General anesthesia

SUMMARY:
Neuromuscular blocking agents are often used during general anesthesia. Also, general anesthesia may be performed without use of neuromuscular blocking agents.

Avoiding neuromuscular relaxation enables better muscle strength recovery.

DETAILED DESCRIPTION:
Rocuronium is well used neuromuscular blocking agent during general anesthesia. Although very often used, neuromuscular blocking agents may sometimes have consequence in form of residual neuromuscular block.

Tha aim of the study is to compare influence of rocuronium during general anesthesia on muscle strength recovery measured by hand grip dynamometer. Measuremwnt of hand grip strength is perforrmed before and after general anesthesia. This research should contribute to better choice of anesthesia technique and better quality of patient recovery, as studies so far have not been detaily carried out.

Hypothesis of the research is that anesthesia without use of neuromuscular blocking agents may enable better recovery of muscle strength in immediate postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* patients ASA status I-III for surgery under general anesthesia
* signed informed consent for participating in research

Exclusion Criteria:

* neuromuscular disease
* poorly controled chronic or acute cardiovascular, respiratory or autoimmune disease
* known allergic reaction to any medication used in this research
* pregnancy
* refusal to participate in this research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Muscle strenght recovery after general anesthesia | Perioperative
  Change in muscle strength recovery measured with hand grip dynamometer after general anesthesia with or without rocuronium. Better understanding of mechanism how neuromuscular blockade influences quality if patient recovery due to muscle strength recovery

CONTACTS AND LOCATIONS:
Locations (1):
- UHCZagreb, Zagreb, Croatia

REFERENCES:
- [Background] Bowman WC. The neuromuscular junction: recent developments. Eur J Anaesthesiol. 1985 Mar;2(1):59-93. No abstract available. PMID 2410263
- [Background] Gatke MR, Viby-Mogensen J, Rosenstock C, Jensen FS, Skovgaard LT. Postoperative muscle paralysis after rocuronium: less residual block when acceleromyography is used. Acta Anaesthesiol Scand. 2002 Feb;46(2):207-13. doi: 10.1034/j.1399-6576.2002.460216.x. PMID 11942873
- [Background] Fuchs-Buder T, Schmartz D. [Residual neuromuscular blockade]. Anaesthesist. 2017 Jun;66(6):465-476. doi: 10.1007/s00101-017-0325-1. German. PMID 28573344